CLINICAL TRIAL: NCT05860699
Title: Cannabidiol as an add-on Treatment During Inpatient Alcohol Cessation in Patients With Severe Alcohol Use Disorder: A Phase II Trial
Brief Title: Cannabidiol as an add-on Treatment During Inpatient Alcohol Cessation : CBD-OH
Acronym: CBD-OH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP180619
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Severe Alcohol Use Disorder (DSM 5)
Keywords: Alcohol use disorder; CBD; Inpatient
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Double Blind Randomized clinical trial with 3 arms :
Who Masked: Outcomes Assessor
Masking Description: Placebo and CBD pills are looking alike and made on purpose for the study by the same manufacturer(Echo Pharmaceutical, BV)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Experimental): add-on placebo (Echo Pharmaceutical, BV) for 11 days during their inpatient stay
  Interventions: Drug: Placebo
- Half-dose CBD (Experimental): add-on cannabidiol (Echo Pharmaceutical, BV) 450 mg per day for 11 days during their inpatient stay
  Interventions: Drug: Half dose CBD
- Full dose CBD (Experimental): add-on cannabidiol (Echo Pharmaceutical, BV) 900 mg per day for 11 days during their inpatient stay
  Interventions: Drug: Full dose CBD

INTERVENTIONS:
Drug: Placebo — Placebo made by the same manufacturer to look like the active pills
  Other Names: Placebo for 11 days during inpatient alcohol cessation
  Arms: Placebo
Drug: Half dose CBD — add-on cannabidiol (Echo Pharmaceutical, BV) 450 mg per day for 11 days during their inpatient stay
  Other Names: Active half-dose for 11 days during inpatient alcohol cessation
  Arms: Half-dose CBD
Drug: Full dose CBD — add-on cannabidiol (Echo Pharmaceutical, BV) 900 mg per day for 11 days during their inpatient stay
  Other Names: Active fulldose of Cannabidiol for 11 days during inpatient alcohol cessation
  Arms: Full dose CBD

SUMMARY:
Randomized clinical trial of 11 days Cannabidiol versus placebo as an adjunctive treatment during inpatient alcohol detoxification to improve abstinence in patients with severe alcohol use disorder.

DETAILED DESCRIPTION:
Primary objective: To increase abstinence maintenance rate at week 6 of the study (1 month after discharge of the scheduled alcohol withdrawal inpatient stay).

Primary Endpoint:

Percentage of patients in each group with documented continuous abstinence at month 1 after discharge, week 6 of the study.

Continuous abstinence will be defined by patient's self-report of alcohol abstinence using standardized TLFB (time line follow back) scales TLFB at screening visit and daily from Day 0 to Day 10 and 4 (1 per week) after discharge up to week 6 of the study) Furthermore, this self-declaration will be confirmed by clinical examination at each study visits assessing acute alcohol intoxication signs and 6 ethyl glucuronide (Et-OH) urinary assessments performed at each study visit (2 during the inpatient stay and 4 (1 per week) after discharge up to week 6 of the study).

Secondary objectives :

* To assess the safety of 11 days of up to 900 mg of cannabidiol as an add-on to usual care in the specific population of patients with severe alcohol use disorder during inpatient alcohol cessation
* In case of relapse, reducing alcohol use after discharge up to week 6 of the study
* To reduce alcohol withdrawal symptoms during inpatient alcohol cessation
* To reduce anxiety symptoms during inpatient alcohol cessation
* In a sub-group of patients: describe CBD plasmatic rate and test if it is correlated with side-effects and/or efficacy
* In the sub-group of patients with co-occuring cannabis use, reducing cannabis use after discharge up to week 6 of the study

Secondary endpoints :

* symptoms check list (PRISE-M) of possible side effects every day from day 1 to 10, and then at each outpatient study visit (4 (1 per week) after discharge up to week 6 of the study). Thus any side effect related to treatment exposure as well as treatment cessation (such as anxiety rebound or withdrawal symptoms related to CBD or increase in cannabis use) could be documented
* in case of relapse: drinking days and drinks per day (self-declared using standardized TLFB time line follow back scale over the past week) at the screening visit and daily from Day 0 to Day 10 and 4 (1 per week) after discharge up to week 6 of the study)
* alcohol withdrawal scales and craving scales (CIWA-R, LIKERT craving scale and an adapt version of the OCDS) at the screening visit and every day from day 0 to 10 then at each study visit: 4 (1 per week) after discharge up to week 6 of the study
* state anxiety scale (STAI-6 the short form of the Spielberger inventory, composed of 6 Likert scales) at the screening visit and every day from day 0 to 10 then at each study visit: 4 (1 per week) after discharge up to week 6 of the study
* Pittsburgh Sleep Quality Index (PSQI) at the screening visit and the last visit. A modified daily version every day from day 0 to 10 then at each study visit a modified weekly version: 4 (1 per week) after discharge up to week 6 of the study
* in the subgroup of patients recruited in Fernand Widal hospital, plasmatic level of CBD will be determined twice: at D5 and D10 of the study by Dr Laurence Labat, head of the toxicology department of Lariboisière hospital. Analysis of cannabinoids in human biological specimens of plasma will rely on an extraction process and a chromatographic separation in LCMSHR (Liquid chromatography coupled to high resolution mass spectrometry) for quantification of Δ9-tetrahydrocannabinol (THC), cannabidiol (CBD), 11-hydroxy Δ9-tetrahydrocannabinol (11-OH THC) and 11-nor-9-carboxy-Δ9-tetrahydrocannabinol (THC-COOH) using deuterated molecules as internal standard. The method was validated in the two biological matrix according to guidelines set forth by COFRAC (Comité d'accréditation Français)
* self-declared current use of all other substances including tobacco products and nicotine replacement therapies, cannabis, and other substances using standardized TLFB (time line follow back) scales ) at the screening visit and every day from day 0 to 10 then at each study visit: 4 (1 per week) after discharge up to week 6 of the study
* in the subgroup of patients who declare themselves as current cannabis users at entry, urinary quantitative determination of cannabinoids by an extraction process and a chromatographic separation in LCMSHR (Liquid chromatography coupled to high resolution mass spectrometry) for quantification of Δ9-tetrahydrocannabinol (THC), cannabidiol (CBD), 11-hydroxy Δ9-tetrahydrocannabinol (11-OH THC) and 11-nor-9-carboxy-Δ9-tetrahydrocannabinol (THC-COOH) using deuterated molecules as internal standard. The method was validated in the two biological matrix according to guidelines set forth by COFRAC (Comité d'accréditation Français). This analyse will be centralized in the toxicology laboratory of Lariboisière hospital (Pr Laurence Labat). This analyse will be performed 6 times: 2 during the inpatient stay (D5 and D10) and 4 (1 per week) after discharge up to week 6 of the study.

DESIGN

Double Blind Randomized clinical trial with 3 arms :

Patients will undergo one or several outpatient screening visits between D-30 and D-1 of inpatient entry.

During this visit, the study design will be fully explained, inclusion and exclusion criteria checked. Patients will be included during this last visit. Three groups of 70 patients each will be randomized 1:1:1 at entry of a scheduled, usually lasting between 11 and 17 days, alcohol inpatient cessation (D0).

They will all receive oxazepam plus an intervention:

* add-on placebo for 11 days during their inpatient stay
* add-on cannabidiol 450 mg per day for 11 days during their inpatient stay
* add-on cannabidiol 900 mg per day for 11 days during their inpatient stay. All groups will undergo the same prospective follow up after discharge with one visit per week to determine if alcohol abstinence is maintained, up to 1-month post-discharge (week 6 of the study).

In case of a relapse, the amount of alcohol used will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for a scheduled alcohol inpatient cessation
* Aged 18-75 years old

  * Meeting DSM 5 criteria for severe AUD
  * Willing to participate
  * Signing a written informed consent
  * Patients with current social insurance
  * For childbearing age, sexually active females: efficacious contraceptive method during treatment and up to seven days after treatment administration

Exclusion Criteria:

* • Patients already scheduled for long term residential care after acute alcohol inpatient detoxification, not able to maintain the outpatient follow up

  * Patients not willing to attend post-discharge visits whatever the reason
  * Any unstable medical condition at entry, such as delirium, acute hepatic failure, hypokalaemia, liver cirrhosis whatever the stage, acute or chronic severe renal failure or any acute psychiatric condition
  * Liver enzymes (ALT and/or AST) above 3 times the upper limit of normal and/or bilirubin above 2 times the upper limit of normal
  * Current medication or need for medication with treatments metabolized by CYP 2C19 or CYP3A4 or UGT enzymes and having strong inhibitor/inducer properties (see list above), and/or current medication or need for medications containing valproate and derivates
  * Any medical history of epileptic seizure
  * Patients with current or past history of cardiac arrhythmias, myocardial infarction and stroke
  * Any history of suicidal attempt in the past 5 years or a score ≥1 to the Suicidal Ideation Attributes Scale (SIDAS)
  * To facilitate efficacy data interpretation, patients currently receiving or wanting to receive another approved pharmacological treatment aimed at alcohol abstinence maintenance (acamprosate, baclofene, disulfiram, nalmefene, naltrexone).
  * Other major current DSM 5 severe substance use disorder (like opiates, cocaine, amphetamines, ...) except for tobacco, cannabis smoking and benzodiazepines use disorders
  * Pregnancy and breast feeding
  * Known hypersensitivity to the active substance or to any of the excipients (including PEG)
  * Patients under guardianship
  * Patients in exclusion periods of other trials
  * Reversely, cannabis use or cannabis use disorders will not be an exclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-05-23 (Estimated); Study Completion 2026-05-23 (Estimated)

PRIMARY OUTCOMES:
clinical abstinence | Week 6
  examination ascertaining documented continuous abstinence (at each study visits assessing acute alcohol intoxication signs) up to month 1 after discharge, week 6 of the study
Self-decalred abstinence verified by the investigator | Week 6
  Self-declared abstinence using standardized TLFB (time line follow back) scales TLFB at screening visit and daily from Day 0 to Day 10 and 4 (1 per week) after discharge up to week 6 of the study).

SECONDARY OUTCOMES:
Biological abstinence | week 6
  6 ethyl glucuronide (EDTA) urinary assessments performed at each study visit (2 during the inpatient stay and 4 (1 per week) after discharge up to week 6 of the study).
Symptoms check list | Day 1 to week 6
  symptoms check list (PRISE-M) of possible side effects every day from day 1 to 10, and then at each outpatient study visit (4 (1 per week) after discharge up to week 6 of the study). Thus any side effect related to treatment exposure as well as treatment cessation (such as anxiety rebound or withdrawal symptoms related to CBD or increase in cannabis use) could be documented
Alcohol reduction in case of relapse | Day 1 to Week 6
  In case of relapse: drinking days and drinks per day (self-declared using standardized TLFB time line follow back scale over the past week) at the screening visit and daily from Day 0 to Day 10 and 4 (1 per week) after discharge up to week 6 of the study)
Reduction of alcohol craving and withdrawal severity | Day 1 to Week 6
  alcohol withdrawal scales and craving scales (CIWA-R, , LIKERT craving scale and an adapt version of the OCDS) at the screening visit and every day from day 0 to 10 then at each study visit: 4 (1 per week) after discharge up to week 6 of the study
Reduction in anxiety | Day 1 to Week 6
  state anxiety scale (STAI-6 the short form of the Spielberger inventory, composed of 6 Likert scales) at the screening visit and every day from day 0 to 10 then at each study visit: 4 (1 per week) after discharge up to week 6 of the study

CONTACTS AND LOCATIONS:
Overall Officials: Florence Vorspan, Principal Investigator — Département de Psychiatrie et de Médecine Addictologique, Hôpital Fernand Widal, AP-HP Inserm UMR-S 1144 Université de Paris FHU NOR-SUD
Locations (12):
- France (12):
  - Hôpital Albert Chenevier, Créteil, Albert Chenevier
  - Hôpital Antoine Béclère, Clamart, Clamart
  - CHU Gabriel Montpied, Clermont-Ferrand, Clermont Ferrand
  - Hôpital Louis Mourier, Colombes, Colombes
  - Hôpital Avicenne, Bobigny, France
  - Hôpital Fernand Widal, Paris, France
  - Hôpital Hôtel-Dieu, Paris, Paris
  - Hôpital Cochin, Paris, Paris
  - Hôpital Saint Anne, Paris, Paris
  - Hôpital Bichat, Paris, Paris
  - Hôpital René Muret, Sevran, Sevran
  - Hôpital la Colombière, Montpellier